CLINICAL TRIAL: NCT04057482
Title: Treatment of Bacterial Vaginosis With Dequalinium Chloride Vaginal Tablets and a Test of Cure Using a New Molecular Diagnostic Test for the Diagnosis of Bacterial Vaginosis
Brief Title: Treatment of BV With Donaxyl and a Molecular Test of Cure
Status: Completed | Type: Observational
Sponsor: Skaraborg Hospital (Other Government)
Responsible Party: Principal Investigator, Per-Goran Larsson, professor, Skaraborg Hospital
Other Study IDs: 2050
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Bacterial Vaginoses
Keywords: Bacterial vaginosis, polymerase chain reaction, molecular diagnostic
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Fumigant 93

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Molecu
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: D — treatment of BV with dequalinium chloride vaginal tablets
  Other Names: dequalinium chloride vaginal tablets

SUMMARY:
. Treatment with dequalinium chloride vaginal tablets for 6 days had a cure rate lower than expected; only 37% of patients were considered cured one month after treatment.

DETAILED DESCRIPTION:
This is the first study to utilize a molecular diagnostic test as a test of cure for bacterial vaginosis. The Nugent score is a reliable method for diagnosing bacterial vaginosis, but similar to traditional clinical diagnostic methods, it is not equally reliable when utilized as a test of cure. This study demonstrated that molecular diagnostic testing can be used as a test of cure and this is the first molecular test that can do that. Treatment with dequalinium chloride vaginal tablets for 6 days had a cure rate lower than expected; only 37% of patients were considered cured one month after treatment.

ELIGIBILITY:
Inclusion Criteria:

BV

Exclusion Criteria:

No other infection (Gc, clhlamydia, trihomonas)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: local maternity and youth clinics in Skaraborg county
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
cure rate of BV | 1 year
  how many that are cured of BV after 1 month

SECONDARY OUTCOMES:
Diagnosis of BV using molecular test | 1 year
  the Kappa index Hay/ison diagnosis and the molecular test

CONTACTS AND LOCATIONS:
Overall Officials: P-G Larsson, PhD, Principal Investigator — överläkare

IPD SHARING:
Plan to Share IPD: No